CLINICAL TRIAL: NCT02524977
Title: Impact of a Quality Improvement And Education Initiative on 'Appropriate' Use of Anticoagulant Therapy in Patients With Atrial Fibrillation
Brief Title: Impact of an Atrial Fibrillation Decision Support Tool (AFDST) on Thromboprophylaxis for Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Pfizer (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Mark Eckman, M.D., Professor of Clinical Medicine, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013-0017; 1UL1TR001425-01 (NIH)
Record Dates: First submitted 2015-08-13; First posted 2015-08-17 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Intervention Only (Active Comparator): Educational Intervention Only - Educational package was delivered as 2 didactic noon-conferences on atrial fibrillation with a review of up-to-date anticoagulation guidelines for stroke prevention, and distribution of educational materials. Physicians delivering the noon conference series at all of the general internal medicine and primary care practice sites included 3 stroke neurologists, 2 cardiologists, and a general internist (PI) who were co-investigators in this study. Internists who were faculty at the University of Cincinnati and Internal Medicine residents also had an opportunity to participate in the first of the noon conferences in a special Department of Medicine Grand Rounds delivered by the PI.
  All practices (intervention and control groups) received the educational package focused on physicians, and clinical and non-clinical staff who would be involved in this QI process.
  Interventions: Behavioral: Educational Intervention Only
- Educational Intervention plus Decision Support (Experimental): Educational Intervention plus Decision Support - Physicians in the intervention arm received a practice-level and physician-level summary report via a secure web site designed for patients with treatment recommendations that were discordant with current therapy, along with an explanation for the recommendation, the gain or loss in QALYs predicted by the decision model and the current 2014 ACC/AHA/HRS guidelines. Providers were also reminded of upcoming visits for patients being seen within the next week so they could review their reports and use them in discussions with their patients.
  Interventions: Behavioral: Decision Support; Behavioral: Educational Intervention Only

INTERVENTIONS:
Behavioral: Decision Support — Provision of recommended antithrombotic therapy based on atrial fibrillation decision support tool that uses both stroke and bleeding risk
  Arms: Educational Intervention plus Decision Support
Behavioral: Educational Intervention Only — Educational conference series

SUMMARY:
Study objective was to improve decision-making and thromboprophylaxis for patients with Atrial Fibrillation (AF) by developing and implementing a computerized decision support tool for individual patient-level decision-making about oral anticoagulant therapy. To accomplish these goals, the investigators studied the incremental impact of adding a quality-improvement (QI) intervention to an educational package (for practice staff and clinicians) using a computerized aid, the Atrial Fibrillation Decision Support Tool (AFDST) for individual patient-level decision-making about oral anticoagulant therapy in patients with non-valvular AF. The decision support tool incorporates individual patients' risk factor profiles for ischemic stroke and bleeding and provides a recommendation for treatment based upon the projected quality-adjusted life expectancy gained or lost with the addition of either oral anticoagulant therapy or aspirin compared with no thromboprophylaxis.

DETAILED DESCRIPTION:
Setting - Cluster randomized trial. Setting - Primary care practices of an integrated healthcare system. Participants - 1,493 adults with non-valvular AF seen between April 2014 and March 2015.

Intervention - Treatment recommendations were made by an Atrial Fibrillation Decision Support Tool (AFDST) based on projections for quality-adjusted life expectancy calculated by a decision analytic model that integrates patient-specific risk factors for stroke and hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects were physicians in our primary care network.
* Patients included in the study were identified through our health system's clinical data store with an International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM), diagnosis of atrial fibrillation (427.31) or atrial flutter (427.32)

Exclusion Criteria:

Diagnoses of mitral valve disease (394.x), aortic valve disease (395.x), heart valve transplant (V42.2) or heart valve replacement (V42.3).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Practices of UC Health, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Eckman MH, Lip GY, Wise RE, Speer B, Sullivan M, Walker N, Kissela B, Flaherty ML, Kleindorfer D, Baker P, Ireton R, Hoskins D, Harnett BM, Aguilar C, Leonard AC, Arduser L, Steen D, Costea A, Kues J. Impact of an Atrial Fibrillation Decision Support Tool on thromboprophylaxis for atrial fibrillation. Am Heart J. 2016 Jun;176:17-27. doi: 10.1016/j.ahj.2016.02.009. Epub 2016 Feb 19. PMID 27264216

RESULTS

PARTICIPANT FLOW:
Groups:
- Educational Intervention Only: Educational Intervention Only - Educational package was delivered as 2 didactic noon-conferences on atrial fibrillation with a review of up-to-date anticoagulation guidelines for stroke prevention, and distribution of educational materials. Physicians delivering the noon conference series at all of the general internal medicine and primary care practice sites included 3 stroke neurologists, 2 cardiologists, and a general internist (PI) who were co-investigators in this study. Internists who were faculty at the University of Cincinnati and Internal Medicine residents also had an opportunity to participate in the first of the noon conferences in a special Department of Medicine Grand Rounds delivered by the PI.
  All practices (intervention and control groups) received the educational package focused on physicians, and clinical and non-clinical staff who would be involved in this QI process.
  Educational Intervention Only: Educational conference series
Period: Overall Study
Arm/Group | Educational Intervention Only | Educational Intervention Plus Decision Support
Started | 738 | 846
Completed | 692 | 801
Not Completed | 46 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Intervention Only | Educational Intervention Plus Decision Support | Total
Number analyzed (Participants) | 692 | 801 | 1493
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean Age | 69.8 (13.5) | 70.2 (13.3) | 70 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 332 | 352 | 684
  Male | 360 | 449 | 809
CHADSVASc [Mean (Standard Deviation); unit: units on a scale] — Scoring Details for CHA2DS2VASc Used to quantify ischemic stroke risk in AF patients.(1) CHA2DS2VASc is an acronym. Each letter stands for a risk factor, assigning 1 point for each of the following: Congestive heart failure, Hypertension, Age 65 - 74, Diabetes, Vascular disease (prior myocardial infarction, peripheral arterial disease, or aortic plaque), and female Sex category. Two points are assigned for a history of Stroke or transient ischemic attack, and Age ≥ 75 years. Score range is 0 - 9. Stroke risk ranges from 0 (for score of zero) to 15.2%/year (for score of 9).
  units on a scale | 3.74 (1.93) | 3.60 (1.86) | 3.67 (1.91)
HAS-BLED [Mean (Standard Deviation); unit: units on a scale] — Scoring Details for HAS-BLED. Used to quantify risk of major bleeding in AF patients receiving treatment with warfarin. HAS-BLED is an acronym. Each letter stands for a risk factor, assigning 1 point for each: poorly controlled Hypertension, Abnormal renal or liver function (one point each), Stroke history, Bleeding history, Labile INR (time in therapeutic range < 60%), Elderly (age ≥ 65), Drugs or alcohol (1 point each - alcohol abuse, or concomitant use of antiplatelet or non-steroidal anti-inflammatory drugs). Risk of major bleeding ranges from 0 (score of 0) to 15.5% (score of 6) per year.
  units on a scale | 2.18 (1.20) | 2.07 (1.15) | 2.12 (1.19)
Proportion Receiving Oral Anticoagulant Therapy [Number; unit: participants] | 346 | 400 | 746

OUTCOME MEASURES:

1. Primary Outcome: Changes in Discordant Antithrombotic Therapy
Description: Changes in the proportion of patients with current therapy that was discordant from the decision support tool recommendation between the start and finish date of the study (one year period).
Time Frame: One year
Population: Patients with an International Classification of Diseases, Ninth Revision, Clinical Modification diagnosis of AF (427.31) or atrial flutter (427.32) who did not have diagnoses of mitral valve disease (394.x), aortic valve disease (395.x), heart valve transplant (V42.2), or heart valve replacement (V42.3) in their active problem list.
Measure: Number; unit: participants
Arm/Group | Educational Intervention Only | Educational Intervention Plus Decision Support
Number analyzed (Participants) | 692 | 801
participants
  Therapy Discordant from AFDST in 2014 | 291 | 335
  Therapy Discordant from AFDST in 2015 | 277 | 329
Statistical Analysis 1: Comparison: Educational Intervention Plus Decision Support; Test type: Superiority or Other; p = 0.02, Chi-squared

2. Secondary Outcome: Antithrombotic Therapy Discordant From AFDST Among Patients for Whom AFDST Report Was Reviewed
Description: Change in discordance between decision support tool recommendation and actual treatment among patients whose physicians reviewed the decision support tool report.
Time Frame: One year
Population: Number of patients for whom antithrombotic therapy was discordant from AFDST recommendation among patients for whom AFDST report was reviewed
Measure: Count of Participants; unit: Participants
Groups:
- 2014: Discordant in 2014
- 2015: Discordant in 2015
Arm/Group | 2014 | 2015
Number analyzed (Participants) | 240 | 240
Participants | 152 | 140

ADVERSE EVENTS:
Arm/Group | Educational Intervention Only | Educational Intervention Plus Decision Support
Serious Adverse Events (participants affected / at risk) | 0/692 | 0/801
Other Adverse Events (participants affected / at risk) | 0/692 | 0/801

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No